CLINICAL TRIAL: NCT07221721
Title: A Pilot Study to Assess the Feasibility and Safety of Targeting Mean Arterial Pressure to Reduce Intra-operative Hypotension
Brief Title: Brain Autoregulation Research Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Marino (Other)
Responsible Party: Sponsor-Investigator, Bradley Marino, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 22-1348
Record Dates: First submitted 2025-10-25; First posted 2025-10-28 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-06

CONDITIONS: Hypotension During Surgery; Hypotension Postprocedural
Keywords: hypotension; neonates; cardiothoracic surgery with cardiopulmonary bypass
MeSH Terms: conditions — Hypotension | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Study) Group (Experimental): Neonates undergoing cardiothoracic surgery (CT) utilizing cardiopulmonary bypass (CPB) who will have active management of their mean arterial pressure (MAP) to keep the MAP above the LLA as measured by a novel autoregulation monitoring modality.
  Interventions: Device: Surgery with Active MAP Management
- Control Group (Sham Comparator): Neonates undergoing cardiothoracic surgery (CT) utilizing cardiopulmonary bypass (CPB) who will have management of their MAP by institutional practice without guidance from an autoregulation monitoring modality.
  Interventions: Other: Surgery without Active MAP Management

INTERVENTIONS:
Device: Surgery with Active MAP Management — Neonates undergoing cardiothoracic surgery (CT) utilizing cardiopulmonary bypass (CPB) who will have active management of their mean arterial pressure (MAP) to keep the MAP above the LLA as measured by a novel autoregulation monitoring modality.
  Arms: Intervention (Study) Group
Other: Surgery without Active MAP Management — Neonates undergoing cardiothoracic surgery (CT) utilizing cardiopulmonary bypass (CPB) who will have management of their MAP by institutional practice without guidance from an autoregulation monitoring modality.
  Arms: Control Group

SUMMARY:
Randomized, multi-site, study assessing the feasibility of lower limit of autoregulation targeted mean arterial pressure (MAP) vs. standard MAP management in neonates undergoing cardiac surgery with cardiopulmonary bypass. After eligibility screening and consent, subjects will be randomized to either the intervention (study) or control group.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is the most common birth defect.1 Surgery to treat CHD is complicated by white matter injury (WMI) on brain magnetic resonance imaging (MRI) and neurodevelopmental (ND) deficits in 50% to 75% of neonates after CHD surgery.2-6 Cerebral hypoperfusion is a major mechanism of brain injury during both cardiopulmonary bypass (CPB) and the perioperative period in the intensive care unit (ICU).7-10 Investigators lack diagnostic and therapeutic means to reduce cerebral hypoperfusion-associated white matter injury (WMI) and improve long-term ND outcomes.11 Our long-term goal is to use real-time measurement of the cerebral lower limit of autoregulation (LLA) to manage arterial blood pressure, reduce cerebral hypoperfusion-associated brain injury, and improve long-term ND outcomes in children at risk for brain hypoperfusion. In a prospective, single blind, randomized clinical trial (RCT) in adults undergoing cardiac surgery, investigators previously showed that targeted LLA arterial blood pressure management to maintain mean arterial pressure (MAP) above the LLA decreased the incidence of postoperative delirium by 45%.12 Our preliminary data indicate that neonates are exposed to significantly more cerebral hypotension than adult patients undergoing CPB. Our central hypothesis is that a strategy of targeting mean arterial pressure (MAP) to a level above an individual's LLA will reduce the risk for WMI and neurodevelopmental impairment in neonates undergoing congenital heart surgery. Our team has validated methodology to delineate the LLA and demonstrated the important role of cerebral autoregulation monitoring on short-term outcomes in CHD subjects who have undergone CPB.13 We can rigorously measure cerebral autoregulation in real time and the amount of cerebral hypotension (duration and magnitude) through the integration of near infrared spectroscopy (NIRS) and the arterial blood pressure.14,15 The efficacy of an LLA targeted MAP strategy to minimize WMI and improve ND outcomes can only be demonstrated by a prospective, single-blind, multi-center randomized RCT. To obtain funding for this large multi-center RCT will require the demonstration of feasibility and safety, as well as, an estimation of the sample size needed to show efficacy.

ELIGIBILITY:
Inclusion Criteria:

* All neonates (<30 days of age)
* Undergoing cardiothoracic surgery with cardiopulmonary bypass

Exclusion Criteria:

* Less than full term (<37 weeks gestation)
* Weight < 2.50kg
* Genetic abnormality or syndrome except heterotaxy syndrome
* Major non-cardiac anomalies (e.g. congenital diaphragmatic hernia, - omphalocele, holoprosencephaly, anencephaly)

Ages: 30 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Hypotension Exposure | From beginning of surgery until 72 hours post-surgery
  Primary outcome is to reduce hypotension exposure, defined as the product of duration and magnitude of arterial blood pressure below LLA measured in the operating room and for the first 72 hours in the ICU.

SECONDARY OUTCOMES:
Aim 2: Lower Limit Autoregulation Monitoring (LLA) | First 30 days post-surgery in the ICU
  To determine LLA targeted MAP vs standard MAP management in real time will not increase perioperative mortality and morbidity in neonates undergoing cardiac surgery with CPB

OTHER OUTCOMES:
Aim 3: Mean Arterial Pressure Management | Seizure assessment by EEG first 48 hours post-op, White matter injury assessment by Brain MRI 7-21 days post-op, neurodevelopmental outcome (neurobehavioral assessment at 30 days or at discharge by the NBO, Bayley-4 at 6 and 12 months).
  Compare LLA targeted MAP vs standard of care MAP management in reducing white matter injury and seizure occurrence and improve neurodevelopment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Marino, MD, MPP, MSSCE, MBA, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No